CLINICAL TRIAL: NCT06797960
Title: ANALGESIC EFFECT of ULTRASOUND GUIDED INTRA- ARTICULAR INJECTION of PLATELET RICH FIBRIN VERSUS INJECTION of HYALURONIC ACID in PATIENTS with MODERATE KNEE OSTEOARTHRITIS. a RANDOMIZED CONTROLLED STUDY
Brief Title: Ultrasound Guided Intra Articular Injection of Platelet Rich Fibrin Versus Hyaluronic Acid As Means of Pain Relief in Patients with Moderate Degree Knee Osteoarthritis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Islam Shaban Shaban, Resident, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: M757
Record Dates: First submitted 2025-01-21; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- PRF group (Active Comparator)
  Interventions: Device: Ultra sound guided Injection of PRF intra articularly
- Hyaluronic acid group (Active Comparator)
  Interventions: Drug: Intra articular injection of HA

INTERVENTIONS:
Device: Ultra sound guided Injection of PRF intra articularly — Intra articular injection of PRF
  Arms: PRF group
Drug: Intra articular injection of HA — Intra articular injection of HA
  Arms: Hyaluronic acid group

SUMMARY:
Randomised controlled trial

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II.
* Moderate knee osteoarthritis

Exclusion Criteria:

* Neurological patients.
* Patients with uncontrolled co morbidities

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pain relief as measured by VAS score | 3 months